CLINICAL TRIAL: NCT03580031
Title: Booster Dose of Human Chorionic Gonadotrophin for Unruptured Follicle in Non IVF/ICSI Cycles: A Randomized Controlled Study
Brief Title: Booster Dose of HCG for Unruptured Follicle in Non IVF/ICSI Cycles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ayman HCG
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: LUF - Luteinised Unruptured Follicle Syndrome
Keywords: LUF; HCG; Booster dose; Ovulation rate; pregnancy rate
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Cohort groups with parallel allocation
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study group (Experimental): HCG IM 10,000 IU Im 48 hours after first triggering dose
  Interventions: Drug: hCG
- Control group (Placebo Comparator): Saline 2m Injection im 48 hours after the first triggering dose
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: hCG — A booster dose (10,000 IU of hCG) was given IM 48 hours after first triggering dose
  Arms: Study group
Drug: Saline Solution — 2 ml of normal saline will be injected 48 hours after first triggering dose
  Arms: Control group

SUMMARY:
This study will be conducted to assess the effect of booster dose of hCG on the unruptured follicles in non IVF/ICSI cycles.

DETAILED DESCRIPTION:
In this study enrolled patients (n=160) who underwent controlled ovarian stimulation and timed intercourse with unruptured mature graffian follicle 48 hours after IM 10,000 IU HCG dose. Patients were allocated randomly into intervention group and control group. In the intervention group another booster dose (10,000 IU of hCG) was given IM while in the control group 2 ml normal saline was given IM leaving follicles for spontaneous rupture

ELIGIBILITY:
Inclusion Criteria:

* Ordinary stimulated cycles
* IUI stimulated cycles
* Unruptured follicle after 10000 IU IM HCG triggering

Exclusion Criteria:

* IVF/ICSI cycles

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Ovulation rate | 48 hours
  rupture of dominant follicle manifested by disappearance of follicle and presence of free fluid in douglas pouch

SECONDARY OUTCOMES:
Pregnancy rate | 15 days
  Number of cases with positive serum pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Dawood, MD, Principal Investigator — Lecturer at Tanta University
Locations (1):
- Ayman Shehata Dawood, Tanta, Algharbia, Egypt

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be displayed